CLINICAL TRIAL: NCT02569242
Title: ONO-4538 Phase III Study A Multicenter, Randomized, Open-label Study in Patients With Esophageal Cancer Refractory or Intolerant to Combination Therapy With Fluoropyrimidine and Platinum-based Drugs
Brief Title: Study of Nivolumab in Unresectable Advanced or Recurrent Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4538-24/CA209-473
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Results first posted 2022-01-14 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-01

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Nivolumab; Docetaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nivolumab Arm (Experimental): Nivolumab 240 mg/body solution intravenously every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Drug: Nivolumab
- Active Comparator Arm （Docetaxel/Paclitaxel） (Active Comparator): Docetaxel: Intravenously administered at a dose of 75 mg/m2 every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  OR
  Paclitaxel: Intravenously administered at a dose of 100 mg/m2 weekly for 6 weeks followed by 2-week drug holiday until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Drug: Docetaxel/Paclitaxel

INTERVENTIONS:
Drug: Nivolumab
  Arms: Nivolumab Arm
Drug: Docetaxel/Paclitaxel
  Arms: Active Comparator Arm （Docetaxel/Paclitaxel）

SUMMARY:
The purpose of study is to evaluate the efficacy and safety of Nivolumab in unresectable advanced or recurrent esophageal cancer patients who have failed in standard chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Men & women ≥20 years of age
* Histologically confirmed unresectable advanced or recurrent esophageal cancer
* Refractory to or intolerant of standard therapy
* ECOG Performance Status score 0 or 1
* A life expectancy of at least 3 months

Exclusion Criteria:

* Current or past history of severe hypersensitivity to any other antibody products
* Patients with multiple primary cancers
* Patients with any metastasis in the brain or meninx that is symptomatic or requires treatment
* Patients with active, known or suspected autoimmune disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharmaceutical Co., Ltd. Ono Pharmaceutical Co., Ltd., Study Director — Ono Pharmaceutical Co. Ltd
Locations (74):
- United States (7):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Georgetown University Med Ctr, Washington D.C., District of Columbia
  - Orlando Health, Inc, Orlando, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke Cancer Institute, Durham, North Carolina
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee
  - The University Of Texas MD Anderson Cancer Center, Houston, Texas
- Odense University Hospital, Odense C, Denmark
- Germany (7):
  - RWTH Aachen University, Aachen
  - Charite Campus Virchow Klinikum, Berlin
  - University Hospital Heidelberg, Heidelberg
  - Universitatsklinikum Jena, Innere Medizin II, Jena
  - MVZ Mitte, Leipzig
  - University Of Mainz Medical Center, Mainz
  - Klinikum reechts der Isar, Technical University Munchen, Munich
- Italy (3):
  - HPG23, Bergamo
  - Fondazione Irccs Istituto Nazionale Tumori, Milan
  - Irccs Istituto Oncologico Veneto Iov, Padua
- Japan (39):
  - Aichi Clinical Site, Nagoya, Aichi-ken
  - Aomori Clinical Site, Hirosaki, Aomori
  - Chiba Clinical Site, Kashiwa, Chiba
  - Ehime Clinical Site, Matsuyama, Ehime
  - Hokkaido Clinical Site, Sapporo, Hokkaido
  - Hyogo Clinical Site, Akashi, Hyōgo
  - Hyogo Clinical Site, Kobe, Hyōgo
  - Kanagawa Clinical Site, Isehara, Kanagawa
  - Kanagawa Clinical Site, Kawasaki, Kanagawa
  - Kanagawa Clinical Site, Yokohama, Kanagawa
  - Mie Clinical Site, Tsu, Mie-ken
  - Miyagi Clinical Site, Sendai, Miyagi
  - Nagano Clinical Site, Saku, Nagano
  - Niigata Clinical Site, Nigatake, Niigata
  - Osaka Clinical Site, Sayama, Osaka
  - Osaka Clinical Site, Suita, Osaka
  - Osaka Clinical Site, Takatsuki, Osaka
  - Saitama Clinical Site, Hidaka, Saitama
  - Saitama Clinical Site, Kita-Adachi County, Saitama
  - Shizuoka Clinical Site, Suntou County, Shizuoka
  - Tochigi Clinical Site, Shimotsuke, Tochigi
  - Tokyo Clinical Site, Bunkyo-ku, Tokyo
  - Tokyo Clinical Site, Chuo-ku, Tokyo
  - Tokyo Clinical Site, Koto-ku, Tokyo
  - Tokyo Clinical Site, Meguro-ku, Tokyo
  - Tokyo Clinical Site, Minato-ku, Tokyo
  - Tokyo Clinical Site, Shinagawa-ku, Tokyo
  - Tokyo Clinical Site, Shinjuku-ku, Tokyo
  - Akita Clinical Site, Akita
  - Chiba Clinical Site, Chiba
  - Fukuoka Clinical Site, Fukuoka
  - Fukushima Clinical Site, Fukushima
  - Hiroshima Clinical Site, Hiroshima
  - Kagoshima Clinical Site, Kagoshima
  - Kumamoto Clinical Site, Kumamoto
  - Kyoto Clinical Site, Kyoto
  - Niigata Clinical Site, Niigata
  - Osaka Clinical Site, Osaka
  - Shizuoka Clinical Site, Shizuoka
- South Korea (7):
  - Busan Clinical Site, Busan
  - Daegu Clinical Site, Daegu
  - Daejeon Clinical Site, Daejeon
  - Gyeonggi-do Clinical Site, Gyeonggi-do
  - Hwasun-Gun Clinical Site, Hwasun-Gun
  - Seoul Clinical Site, Seoul
  - Ulsan Clinical Site, Ulsan
- Taiwan (8):
  - Changhua Clinical Site, Changhua
  - Chiayi Clinical Site, Chiayi City
  - Kaohsiung Clinical Site, Kaohsiung City
  - Keelung Clinical Site, Keelung
  - Taichung Clinical Site, Taichung
  - Tainan Clinical Site, Tainan
  - Taipei Clinical Site, Taipei
  - Taoyuan Clinical Site, Taoyuan District
- United Kingdom (2):
  - Velindre Cancer Centre, Cardiff, Cardiganshire
  - The Beatson West Of Scotland Cancer Centre, Glasgow, Lanarkshire

IPD SHARING:
Plan to Share IPD: Yes
URL: https://www.ono.co.jp/eng/rd/policy.html

REFERENCES:
- [Derived] Kato K, Cho BC, Takahashi M, Okada M, Lin CY, Chin K, Kadowaki S, Ahn MJ, Hamamoto Y, Doki Y, Yen CC, Kubota Y, Kim SB, Hsu CH, Holtved E, Xynos I, Kodani M, Kitagawa Y. Nivolumab versus chemotherapy in patients with advanced oesophageal squamous cell carcinoma refractory or intolerant to previous chemotherapy (ATTRACTION-3): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2019 Nov;20(11):1506-1517. doi: 10.1016/S1470-2045(19)30626-6. Epub 2019 Sep 30. PMID 31582355

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator Arm （Docetaxel/Paclitaxel）: Docetaxel: Intravenously administered at a dose of 75 mg/m2 every 3 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  OR
  Paclitaxel: Intravenously administered at a dose of 100 mg/m2 weekly for 6 weeks followed by 2-week drug holiday until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
Period: Overall Study
Arm/Group | Nivolumab Arm | Active Comparator Arm （Docetaxel/Paclitaxel）
Started (Enrolled and randomly assigned) | 210 (Included in intention-to-treat analysis for overall survival and progression-free survival) | 209 (Included in intention-to-treat analysis for overall survival and progression-free survival)
Completed (Received assigned treatment of IMP) | 209 (Analysed for safety) | 208 (Analysed for safety)
Not Completed | 1 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab Arm | Active Comparator Arm （Docetaxel/Paclitaxel） | Total
Number analyzed (Participants) | 210 | 209 | 419
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 112 | 85 | 197
  >=65 years | 98 | 124 | 222
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 64 [57 to 69] | 67 [57 to 72] | 65 [57 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 24 | 55
  Male | 179 | 185 | 364
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 201 | 200 | 401
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 201 | 200 | 401
  White | 9 | 9 | 18
ECOG performance status [Count of Participants; unit: Participants] — performance status 0；Fully active, able to continue all pre-disease activities without restriction performance status 1；Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work
  Participants
    0 | 101 | 107 | 208
    1 | 109 | 102 | 211
Disease stage : TNM classification [Count of Participants; unit: Participants] — In this study, the TNM Classification of Malignant Tumours, Seventh Edition, published by the Union for International Cancer Control (UICC) (hereinafter referred to as "the TNM classification") will be used to determine disease stage. please refer to the protocol information. Higher numbers mean the cancer is more advanced. Population: Summarized for subjects with non-recurrent esophageal cancer.
  Participants
    II - III: number analyzed (Participants) | 107 | 120 | 227
    II - III | 8 | 13 | 21
    IV: number analyzed (Participants) | 107 | 120 | 227
    IV | 94 | 100 | 194
    unknown: number analyzed (Participants) | 107 | 120 | 227
    unknown | 5 | 7 | 12
Previous therapies [Count of Participants; unit: Participants]
  Surgery | 111 | 94 | 205
  Radiothrapy | 153 | 142 | 295
  Systemic anticancer therapy | 210 | 208 | 418
Number of organs of metastases [Count of Participants; unit: Participants]
  <=1 | 89 | 91 | 180
  >=2 | 121 | 118 | 239
Site of metastases [Count of Participants; unit: Participants]
  Lymph node | 159 | 163 | 322
  Liver | 57 | 54 | 111
  Lung | 98 | 92 | 190
  Bone | 23 | 25 | 48
PD-L1 expression [Count of Participants; unit: Participants] — In this study, the subject will test positive for PD-L1 when cancerous cells with stained cell membranes account for ≧1% of at least 100 evaluable cancerous cells and will test negative for PD-L1 when such cells account for <1%, the same applies to 5% and 10%.
  Participants
    <1% | 109 | 107 | 216
    >=1% | 101 | 102 | 203
    <5% | 136 | 137 | 273
    >=5% | 74 | 72 | 146
    <10% | 146 | 152 | 298
    >=10% | 64 | 57 | 121
History of smoking [Count of Participants; unit: Participants]
  Never | 30 | 32 | 62
  Former | 159 | 147 | 306
  Current | 21 | 30 | 51

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: ("Date of death from any cause" - "Date of randomization" + 1) / 30.4375. For subjects lost to follow-up and subjects who are alive at the time of data cutoff date, data will be censored at the time the subject was last confirmed to be alive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Arm | Active Comparator Arm （Docetaxel/Paclitaxel）
Number analyzed (Participants) | 210 | 209
months | 10.9 [9.2 to 13.3] | 8.4 [7.2 to 9.9]

2. Secondary Outcome: Progression-free Survival
Description: Please refer to the protocol, overall response and best overall response will be determined solely by imaging assessment according to the RECIST Guideline Version 1.1, and will not take into account any clinical/symptomatic progression. Evaluable imaging data will be overall response without an overall response of "Not Evaluable (NE)."
Time Frame: ("Earlier date on which either the overall response was assessed as PD or the subject died of any cause" - "Date of randomization" + 1) / 30.4375.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Arm | Active Comparator Arm （Docetaxel/Paclitaxel）
Number analyzed (Participants) | 210 | 209
months | 1.7 [1.5 to 2.7] | 3.4 [3.0 to 4.2]

3. Secondary Outcome: Duration of Response
Description: as for outcome 2
Time Frame: ("Earlier date on which either the overall response was assessed as PD for the first time after confirmed response or the subject died of any cause" - "Date of first assessment of confirmed CR or PR" + 1) / 30.4375.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Arm | Active Comparator Arm （Docetaxel/Paclitaxel）
Number analyzed (Participants) | 210 | 209
months | 6.9 [5.4 to 11.1] | 3.9 [2.8 to 4.2]

ADVERSE EVENTS:
Time Frame: Monitoring for any AEs will be continued until 28 days after the end of the treatment phase. In subjects who, at the time of initiation of the follow-up investigation, have any AE for which a causal relationship to the investigational product cannot be ruled out or which led to discontinuation, investigation of the AE will be continued until the event is judged not to require further follow-up. SAEs are to be collected during the treatment period and for 100 days following the last dose.
Description: For all-cause mortality, the number of adverse events reported as Grade 5 was extracted.
Arm/Group | Nivolumab Arm | Active Comparator Arm （Docetaxel/Paclitaxel）
All-Cause Mortality (participants affected / at risk) | 7/209 | 5/208
Serious Adverse Events (participants affected / at risk) | 68/209 | 77/208
Other Adverse Events (participants affected / at risk) | 185/209 | 204/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Arm (N=209) | Active Comparator Arm （Docetaxel/Paclitaxel） (N=208)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 16
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Gastric fistula (Gastrointestinal disorders) | 1 | 0
Aorto-oesophageal fistula (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 1
Pyrexia (General disorders) | 6 | 1
Sudden death (General disorders) | 1 | 1
Disease progression (General disorders) | 0 | 1
Stenosis (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 2
Mediastinitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 10 | 13
Postoperative wound infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Anal abscess (Infections and infestations) | 0 | 1
Muscle abscess (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 1 | 5
Infectious pleural effusion (Infections and infestations) | 0 | 2
Spinal cord abscess (Infections and infestations) | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Stoma site extravasation (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 3
Liver function test increased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 6
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Jejunostomy (Surgical and medical procedures) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Arm (N=209) | Active Comparator Arm （Docetaxel/Paclitaxel） (N=208)
Anaemia (Blood and lymphatic system disorders) | 24 | 61
Leukopenia (Blood and lymphatic system disorders) | 0 | 18
Neutropenia (Blood and lymphatic system disorders) | 1 | 40
Hypothyroidism (Endocrine disorders) | 21 | 3
Abdominal pain (Gastrointestinal disorders) | 12 | 8
Constipation (Gastrointestinal disorders) | 35 | 40
Diarrhoea (Gastrointestinal disorders) | 36 | 34
Dysphagia (Gastrointestinal disorders) | 13 | 3
Nausea (Gastrointestinal disorders) | 23 | 40
Stomatitis (Gastrointestinal disorders) | 7 | 26
Vomiting (Gastrointestinal disorders) | 12 | 17
Chest pain (General disorders) | 13 | 4
Fatigue (General disorders) | 19 | 52
Malaise (General disorders) | 12 | 49
Pyrexia (General disorders) | 29 | 38
Nasopharyngitis (Infections and infestations) | 13 | 9
Upper respiratory tract infection (Infections and infestations) | 15 | 13
Alanine aminotransferase increased (Investigations) | 11 | 7
Aspartate aminotransferase increased (Investigations) | 13 | 7
Lymphocyte count decreased (Investigations) | 5 | 21
Neutrophil count decreased (Investigations) | 3 | 76
Weight decreased (Investigations) | 11 | 11
White blood cell count decreased (Investigations) | 2 | 72
Decreased appetite (Metabolism and nutrition disorders) | 40 | 68
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 22
Dysgeusia (Nervous system disorders) | 5 | 14
Neuropathy peripheral (Nervous system disorders) | 0 | 23
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 48
Insomnia (Psychiatric disorders) | 11 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 100
Pruritus (Skin and subcutaneous tissue disorders) | 26 | 15
Rash (Skin and subcutaneous tissue disorders) | 26 | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT02569242/Prot_SAP_000.pdf